CLINICAL TRIAL: NCT03206372
Title: Risk of Venous Thromboembolism in First Degree Relatives of Women With or Without Venous Thromboembolism During Hormonal Exposure
Brief Title: Risk Factors of Venous Thromboembolism in Women During Hormonal Exposure
Acronym: FIT-H
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: FIT-H (29BRC17.0063)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolic Disease
MeSH Terms: interventions — Diagnosis-Related Groups; Control Groups

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — frozen plasma for DNA analysis (Factor V Leiden and prothrombin gene mutation) stored in central lab in Brest at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: The cases are the first-degree family members of propositi having had an thromboembolic venous disease in hormonal context.
  Interventions: Other: Case group
- Control group: The controls are the first-degree family members of propositi who have never had an thromboembolic venous disease and have identical hormonal exposure
  Interventions: Other: Control group

INTERVENTIONS:
Other: Case group — Questionnaire to be completed, blood sample and possibly echo-doppler
  Groups: Case group
Other: Control group — Questionnaire to be completed, blood sample and possibly echo-doppler
  Groups: Control group

SUMMARY:
Young women have an increased risk of venous thromboembolism (VTE) during hormonale exposure (estrogen-containing pill or pregnancy). In order to detect women at higher risk of VTE during hormonal exposure, thrombophilia testing is often performed in order to adapt contraception methods and/or to increases thromboprophylaxy during pregnancy. However, such practice is probably not accurate nor discriminent. Indeed, there are evidence that the impact of the familial history of VTE might be stronger than that of detectable inherited thrombophilia.

The "FIT-H" study is a cross-sectional study comparing the prevalence of previous venous thromboembolism in first-degree relatives of women (propositi) who had a first episode of venous thromboembolism in association with hormonal exposure with the prevalence of previous venous thromboembolism in first-degree relatives of women who did not have venous thromboembolism during a similar hormonal exposure.

The primary objective is to determine the association between the presence or the absence of VTE in young women during hormonal exposure and the presence or the absence of a previous episode of VTE in their first-degree relatives. Secondary objective is to determine the impact of associated inherited thrombophilia on the risk of VTE in first-degree relatives.

DETAILED DESCRIPTION:
Rational

The annual incidence of venous thromboembolism (VTE) is about 1 to 2/1000 person-years and mortality is 10% when VTE occurs as pulmonary embolism. VTE is a multifactorial disease caused by hereditary and acquired risk factors. Among the latter, hormonal exposure in young women (estrogen-containing pill, pregnancy) remains a major health issue given the frequency of this condition and the 4 to 5-fold increased risk of VTE in the presence of such exposure. In practice, inherited thrombophilia screening is often performed with the aim to identify young women at higher risk for VTE and to avoid estrogen-containing pill or to reinforce thromboprophylaxis during pregnancy. The increased risk of thrombosis in relatives is incompletely explained by the presence of known thrombophilias, as the risk of thrombosis in first-degree relatives is increased even if patients do not have a detectable defect.

In a large cross-sectional study including 2830 first-degree relatives of patients with VTE, we previously showed that the risk of VTE in the first-degree relatives of patients with a first VTE is strongly influenced by whether the VTE was provoked or unprovoked, the patient's age when the VTE occurred, and the number of relatives who have had thrombosis. The risk of VTE in first-degree relatives is about twice as high if the index case had an unprovoked compared to a provoked VTE, is about three times as high if the index case had VTE before about 50 years compared to later in life, and at least twice as high if two rather than one family members have had VTE. The influence of these factors on the risk of VTE in first-degree relatives was additive, and occurred independently of the presence of factor V Leiden or the prothrombin 20210A gene in index cases.

The underlying hypothesis is that patients who have unprovoked VTE or at a young age often have undetected hereditary thrombophilias and that these defects increase the risk of thrombosis in their relatives. However, the number of included young women in the study was to low to confirm if such familial risk was also elevated if young women were on hormonal exposure.

In the present study, our hypothesis is that the risk of VTE in first-degree relatives of young women with VTE on hormonal exposure will be higher than that in first-degree relatives of young women on a similar hormonal exposure without VTE, independently of the presence or not of a detectable inherited thrombophilia.

Methods

Design: French multicentre prospective cross-sectional case-control study comparing the prevalence of VTE in first-degree relatives (subjects) of young women with VTE during hormonal exposure (propositus) with the prevalence of VTE in first-degree relatives (subjects) of young women without VTE during a similar hormonal exposure (propositus).

Objectives

* Primary objective: to demonstrate that 1st-degree relatives (study subjects) of patients of childbearing age (propositi) with a first episode of MVTE in a hormonal context* have a higher risk of MTVE than 1st-degree relatives of propositi exposed to the same hormonal context and without MVTE.
* Secondary objectives:

  1. determine the association between family risk of VTE and the presence, in the propositi, of a frequent hereditary thrombophilia (factor V Leiden, G20210A mutation of the prothrombin gene);
  2. determine the impact of other variables on family risk of VTE: (age at onset of VTE, severity of VTE, number of symptomatic family members).

     Primary outcome: the presence of symptomatic VTE in 1st-degree relatives.

     Study population

     Eligibility criteria:
* Propositi with objectively confirmed proximal deep vein thrombosis (i.e. ultrasonography) or pulmonary embolism (i.e. lung scanning) in women (18 to 50 years) while on hormonal exposure.

Inclusion criteria

* First-degree relatives (biological parents, brothers, sisters, children) of women of childbearing age 18 to 50 years (propositus) with a first MVTE in the hormonal setting and matched control women in the same hormonal setting who have never had MVTE, consenting to first-degree relatives being contacted to participate in the present study.
* Written consent from propositi and family members.

Exclusion criteria

* First-degree relatives whose propositus received preventive antithrombotic medication during pregnancy or contraception.
* Family members of propositus who have had superficial or muscular venous thrombosis
* No information can be obtained on first-degree relatives.
* Family members under 16 years of age.
* Vulnerable persons other than minors aged 16 to 18 (guardianship, curatorship).
* Non-affiliated and non-beneficiary of a health insurance scheme.

Matching criteria

First degree relatives "cases" will matched (1:1) with first-degree relatives "controls" via their propositi characteristics based on the following keys:

* age ±2 years
* hormonal exposure (pregnancy or estrogen-containing pill)
* tobacco smoking
* BMI

Previous VTE in First-Degree Relatives

* Using a previously described algorithm, first-degree relatives were classified as "have had VTE" if they satisfied either of the following two criteria. First, results of diagnostic testing were available that documented previous deep vein thrombosis (including thrombosis confined to the distal deep veins) or pulmonary embolism. Second, they had, in addition to a history of symptoms suggestive of VTE, at least one of the following: i) a history of having been treated with anticoagulant therapy for at least two months without another indication; or ii) a current ultrasound examination that showed that the proximal deep veins were not fully compressible or that there was reflux in a popliteal vein; or iii) current symptoms and signs suggestive of the post-thrombotic syndrome (defined as a score ≥5 on the Villalta scale).
* Relatives were classified as "have not had VTE" if they satisfied all of the following criteria: 1) no known or suspected previous diagnosis of VTE; and 2) no unexplained anticoagulation in the past; and 3) did not currently have symptoms or signs suggestive of the post thrombotic syndrome (i.e., had a score <5 on the Villalta scale).
* Relatives were classified as "uncertain for previous VTE" if they did not satisfy the criteria for either previous, or no previous, VTE.

Factor V Leiden and the Prothrombin 20210A Gene Variant After first-degree relatives had completed assessments for previous VTE, their index cases will categorized as positive for factor V Leiden or the prothrombin 20210A gene variant, or negative for both. Personnel who will be unaware of the propositus family history of VTE, or the subject's past history of VTE, will perfome these assays in a central laboratory in France.

ELIGIBILITY:
Eligibility criteria:

- Propositi with objectively confirmed proximal deep vein thrombosis (i.e. ultrasonography) or pulmonary embolism (i.e. lung scanning) in women (18 to 50 years) while on hormonal exposure.

Inclusion criteria

* First-degree relatives (biological parents, brothers, sisters, children) of women of childbearing age 18-50 years (propositus) with a first MVTE in the hormonal setting and matched control women in the same hormonal setting who have never had MVTE, consenting to first-degree relatives being contacted to participate in the present study.
* Written consent from propositi and family members.

Exclusion criteria

* First-degree relatives whose propositus received preventive antithrombotic medication during pregnancy or contraception.
* Family members of propositus who have had superficial or muscular venous thrombosis
* No information can be obtained on first-degree relatives.
* Family members under 16 years of age.
* Vulnerable persons other than minors aged 16 to 18 (guardianship, curatorship).
* Not affiliated to or not benefiting from a health insurance scheme.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Definitions
  * cases are first-degree relatives (i.e., parents, siblings, children) of young women who have VTE during hormonal exposure;
  * controls are first-degree relatives (i.e., parents, siblings, children) of young women who did not have VTE during a similar hormonal exposure;
  * study subjects are first-degree relatives
  * propositi are young women on hormonal exposure, whether VTE was present of not
  * hormonal exposure is defined by estrogen-containg pill exposure (ongoing or stopped from less than 3 months) or pregnancy or post-partum (in the three months following delivery), in the absence of other provoking risk factors (such as surgery, prolonged immobilization or trauma of lower limbs in the past three months, or cancer in the past 2 years)
Sampling Method: Non-Probability Sample
Enrollment: 2640 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Presence of venous thromboembolic disease in first-degree relatives. | 1 day
  The primary outcome measure is defined by the presence of symptomatic venous thromboembolic disease in first degree relatives based on:
  * objective, validated and standardized criteria
  * or a validated and standardized questionnaire and leg ultrasound according to a validated algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Francis Couturaud, MD, PhD, Principal Investigator — EA3878 (GETBO), Brest University Hospital in France
Locations (8):
- France (8):
  - CHRU Brest, Brest
  - HIA, Brest
  - Clermont Ferrand, Clermont-Ferrand
  - CH Morlaix, Morlaix
  - Paris HEGP, Paris
  - RENNES, Rennes
  - Saint Etienne, Saint-Etienne
  - Tours, Tours

IPD SHARING:
Plan to Share IPD: No